CLINICAL TRIAL: NCT05945225
Title: Clinical Comparison of Two Sonic Electric Toothbrushes and Two Manual Toothbrushes, Used Under Normal Oral Hygiene Conditions, on the Reduction of Gingival Inflammation in Pregnant Women Aged 18 to 40: Randomized Clinical Trial
Brief Title: Pregnancy Women and Individual Oral Prophylaxis in the Control of Gingival Inflammation (PRE-IOP)
Acronym: PRE-IOP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Collaborators: University of Nancy (Other); Elsan (Other)
Responsible Party: Principal Investigator, Carrouel Florence, Associate professor, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRE-IOP
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pregnant Woman
Keywords: manual toothbrush; electric sonic toothbrush; oral prophylaxis; pregnant woman; gingival inflammation
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group using sonic toothbrush (Experimental): Patient will be asked to use a sonic toothbrush for 3 months
  Interventions: Device: Sonicare DiamondClean 9000 Philips®
- Group using hydrosonic toothbrush (Experimental): Patient will be asked to use a hydrosonic toothbrush for 3 months
  Interventions: Device: HydroSonic Easy Curaden®
- Group using manual toothbrush with 5460 strands (Experimental): Patients will be asked to use a manual toothbrush with 5460 strands for 3 months
  Interventions: Device: Manual toothbrush Curaprox CS 5460
- Group using manual toothbrush (Placebo Comparator): Patients will be asked to use a manual toothbrush for 3 months
  Interventions: Device: Manual toothbrush Oral-B 123

INTERVENTIONS:
Device: Sonicare DiamondClean 9000 Philips® — Brush teeth with the electric toothbrush daily during 3 months
  Arms: Group using sonic toothbrush
Device: HydroSonic Easy Curaden® — Brush teeth with the hydrosonic toothbrush daily during 3 months
  Arms: Group using hydrosonic toothbrush
Device: Manual toothbrush Oral-B 123 — Brush teeth with the manual toothbrush daily during 3 months
  Arms: Group using manual toothbrush
Device: Manual toothbrush Curaprox CS 5460 — Brush teeth with the manual toothbrush daily during 3 months
  Arms: Group using manual toothbrush with 5460 strands

SUMMARY:
Gingivitis in pregnant women is a common inflammatory periodontal disease that appears from the third month of pregnancy with an overall prevalence of 35 to 100%. This condition is induced by oral biofilm and exacerbated by increased levels of sex steroid hormones characteristic of pregnancy. Strict bacterial plaque control with both professional and home oral hygiene is essential. Manual toothbrushes require a more specific manual technique for women, while sonic electric toothbrushes, due to their ease of use, might be an excellent for oral individual prophylaxis. Therefore, the question of which type of manual or electric toothbrush might be more effective in reducing gingival inflammation in pregnant women is still unresolved. In literature there are a large number of in vitro clinical studies on this topic, there are currently no clinical studies investigating this long-term clinical comparison.

In this context, this study is a randomized clinical trial consisting of a comparative evaluation between two manual and two sonic electric toothbrushes in the efficacy of the control of plaque in order to reduce gingivitis in women during the period of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 40 years of age
* 15-18 weeks pregnant
* Acceptance of study terms and conditions
* Signature of informed consent form

Exclusion Criteria:

* Protected women
* Stage II,III periodontal disease (i.e. PD ≥ 4 mm, and/or CAL ≥ 4 mm), generalized (>30% od sites)
* History or treatment of periodontal disease
* Current dental or orthodontic treatment
* Fewer than 20 natural teeth, excluding third molars
* Taking medication affecting the gums and/or oral mucosa
* Regular use (more than once a week) of interdental brushes and/or dental floss and/or mouthwash
* Removable prosthesis
* Dental implants
* Systemic disorder such as blood disorders, diabetes, and risk of endocarditis infections
* Anticoagulant treatment
* Inability to follow protocol or non-cooperation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 120 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of gingival bleeding from baseline during woman pregnancy | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  Change of gingival inflammation in pregnant woman using manual or electric toothbrushes in daily practice

SECONDARY OUTCOMES:
Effect on gingival bleeding | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  Bleeding on Probing
Effect on gingival inflammation | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  gingival index
Effect on dental plaque | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  plaque index
Effect on gingival attachment | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  clinical attachment loss
Effect on Periodontal Pocket | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  Periodontal Pocket Probing Depth
Customer Satisfaction Score | T1 (Baseline), T2 (+ 1 month) and T3 (+ 3 months)
  * the minimum and maximum values: 1, 7
  * lower scores mean a worse outcome.
  * the minimum and maximum values: 1, 7
  * lower scores mean a worse outcome.
  * the minimum and maximum values: 1, 7
  * lower scores mean a worse outcome. The score range from 1 (minimum) to 7 (maximum). Lower score mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Majorelle, Nancy, France

IPD SHARING:
Plan to Share IPD: No